CLINICAL TRIAL: NCT03750799
Title: Cross-training Effect of Whole-body Vibration
Acronym: CTEWBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan KARACAN, Researcher, Assoc Prof, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IstPMRTRH-BMR2
Record Dates: First submitted 2018-11-18; First posted 2018-11-23 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Muscle Physiology

STUDY DESIGN:
Intervention Model Description: Experimental group was exposed WBV, Control group was exposed sham WBV
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All of the participants were told that the vibration stimulation was performed for muscle strengthening. However, participants had no knowledge about the characteristics of the vibration used for muscle-strength enhancement. Vibration was applied in the experimental group, whereas sham vibration was applied in the Control group. The WBV exercise was performed at different days for the Control and Experimental groups to make them blind to each other's applications.All measurements were made by an independent assessor (isokinetic test laboratory assistant) blinded to the trial allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Whole body vibration was applied on the right lower extremity.
  Interventions: Device: Whole body vibration
- Sham group (Sham Comparator): Unlike the experimental group, sham vibration was applied to the control group.
  Interventions: Device: Sham vibration

INTERVENTIONS:
Device: Whole body vibration — Whole body vibration was applied on the right lower extremity in the experimental group.
  Arms: Experimental group
Device: Sham vibration — Sham vibration was applied on the right lower extremity in the Control sham group
  Arms: Sham group

SUMMARY:
This study evaluates whether an increase in the ipsilateral knee flexor muscle strength transfers to the contralateral knee extensors which are not exposed to vibration, when unilateral-isolated whole body vibration (WBV) is applied to the lower extremity. In the half of volunteers the right leg were exposed vibration, while in the other half the right leg were exposed sham vibration. Muscle strength were measured with the Cybex® (Massachusetts, USA) extremity-testing system.

DETAILED DESCRIPTION:
This study was included 40 healthy volunteers. The change in the quadriceps muscle strength after 20 session of WBV exercises was evaluated this study. In the WBV group, 20 sessions of unilateral lower extremity vibration exercises were performed with the Whole Body Vibration (WBV) device. WBV was applied when the subjects are in the semi-squat position. WBV was implemented with Powerplate® Pro5 (PowerPlate® International Ltd, London, United Kingdom). During 20 sessions, the WBV amplitude and vibration time were increased gradually. In the first session, the subjects were do a 30-second, 30-35, 40- and 45-Hz low-amplitude WBV while the knee and hip joint were in 30 degrees of flexion (in the semi-squat position); 10-second rest period between vibration applications were applied. A total duration of WBV was be two minutes. In the 20th session, the subjects were given a 60-second, 30-, 35-, 40- and 45-Hz high-amplitude WBV while the knee and hip joint were in 45 degrees of flexion; 10-second rest period between vibration applications were applied. A total duration of WBV was eight minutes. During WBV, the left lower extremity was in the knee-hip flexion position but was not exposed the vibration.

The same experimental protocol was applied to the isometric exercise (control) group. Unlike the experimental group, sham vibration was applied to the control group. Before and after 20 session-exercise, both knee extensor isokinetic muscle strength was measured.

ELIGIBILITY:
Inclusion Criteria:

* Men with ages between 20-50 years
* Being healthy
* Being volunteer
* Right-sided dominant

Exclusion Criteria:

* Non-cooperative subject

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Muscle strength gain of the untrained contralateral quadriceps muscle | four months
  Untrained contralateral quadriceps muscle strength was measured with the Cybex extremity-testing system before and after trial. Unit of this parameter was Nm

CONTACTS AND LOCATIONS:
Overall Officials: Ilhan Karacan, Assoc Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karacan I, Cidem M, Cidem M, Turker KS. Whole-body vibration induces distinct reflex patterns in human soleus muscle. J Electromyogr Kinesiol. 2017 Jun;34:93-101. doi: 10.1016/j.jelekin.2017.04.007. Epub 2017 Apr 24. PMID 28457998
- [Background] Karacan I, Cidem M, Yilmaz G, Sebik O, Cakar HI, Turker KS. Tendon reflex is suppressed during whole-body vibration. J Electromyogr Kinesiol. 2016 Oct;30:191-5. doi: 10.1016/j.jelekin.2016.07.008. Epub 2016 Jul 25. PMID 27485766
- [Background] Cakar HI, Cidem M, Sebik O, Yilmaz G, Karamehmetoglu SS, Kara S, Karacan I, Turker KS. Whole-body vibration-induced muscular reflex: Is it a stretch-induced reflex? J Phys Ther Sci. 2015 Jul;27(7):2279-84. doi: 10.1589/jpts.27.2279. Epub 2015 Jul 22. PMID 26310784
- [Background] Karamehmetoglu SS, Karacan I, Cidem M, Kucuk SH, Ekmekci H, Bahadir C. Effects of osteocytes on vibration-induced reflex muscle activity in postmenopausal women. Turk J Med Sci. 2014;44(4):630-8. PMID 25551934
- [Background] Cidem M, Karacan I, Diracoglu D, Yildiz A, Kucuk SH, Uludag M, Gun K, Ozkaya M, Karamehmetoglu SS. A Randomized Trial on the Effect of Bone Tissue on Vibration-induced Muscle Strength Gain and Vibration-induced Reflex Muscle Activity. Balkan Med J. 2014 Mar;31(1):11-22. doi: 10.5152/balkanmedj.2013.9482. Epub 2014 Mar 1. PMID 25207162
- [Background] Cakar HI, Cidem M, Kara S, Karacan I. Vibration paradox and H-reflex suppression: is H-reflex suppression results from distorting effect of vibration? J Musculoskelet Neuronal Interact. 2014 Sep;14(3):318-24. PMID 25198227